CLINICAL TRIAL: NCT04385212
Title: COVIDAge Study- Hospital Des Trois-Chêne
Brief Title: Outcomes in Hospitalized Older Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Christine Serratrice, MD, Principal Investigator, University Hospital, Geneva
Other Study IDs: 2020-00819
Record Dates: First submitted 2020-04-29; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus Infection; Sars-CoV2; Elderly Infection; Old Age; Debility
MeSH Terms: conditions — Coronavirus Infections; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In December 2019, the first patients infected with the 2019 novel coronavirus (2019-nCoV) were diagnosed in Wuhan. The clinical presentation and course of Severe Acute Respiratory Syndrome-CoV-2 (SARS-CoV-2) infection is poorly understood in older patients and is certainly different from the general population. This project is designed to better understand and to determine clinical, biological and radiological markers of poor adverse outcomes in hospitalized older patients diagnosed with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19, defined by a positive polymerase chain reaction (PCR) test for SARS-CoV-2 detection, obtained by a nasopharyngeal swab or sputum sample.
* Or patients with negative virus detection in the PCR test, but with a high clinical suspicion will also be considered with COVID-19.

Exclusion Criteria:

- Presence of document indicating a refusal to participate in a research study.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: All the patients hospitalized in our geriatrics department with Sars-Cov-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
To evaluate the relative contributions of comorbidities on intra-hospitalized death | 1 month
  We measure functional score of comorbidities

SECONDARY OUTCOMES:
To evaluate the relative contributions of functional characteristics on intra-hospitalized death | 1 month
  We measure Functional Independence Measure scale
To explore specific clinical profiles that may influence COVID-19 disease outcomes in the elderly based on geriatrics syndromes | 1 month
  We describe the role fo geriatric syndrome such as delirium, falls

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation and Geriatrics, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided